CLINICAL TRIAL: NCT00069329
Title: A Long-Term Outcome Study With the IL-1 Receptor Antagonist Anakinra/Kineret in Patients With Neonatal Onset Multisystem Inflammatory Disease (NOMID/CINCA Syndrome) A Therapeutic Approach to Study the Pathogenesis of This Disease
Brief Title: Anakinra to Treat Patients With Neonatal Onset Multisystem Inflammatory Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: data submitted for Food and Drug Administration (FDA) approval
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 030298; ZIAAR041138-08 (NIH); NCT00069329 (Other: National Institutes of Health); 03-AR-0298 (Other: NIHCC)
Record Dates: First submitted 2003-09-22; First posted 2003-09-23 (Estimated); Results first posted 2016-12-01 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-10

CONDITIONS: Nervous System Malformations; Arthropathy, Neurogenic; Urticaria; Papilledema
Keywords: Central Nervous System; Abnormalities; Arthropathy; Urticaria; Papilledema; Auto-Inflammation; Inflammatory Disease; Neonatal Onset Multisystem Inflammatory Disease; NOMID; CINCA Syndrome
MeSH Terms: conditions — Nervous System Malformations; Arthropathy, Neurogenic; Urticaria; Papilledema; Congenital Abnormalities; Joint Diseases; Cryopyrin-Associated Periodic Syndromes | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NOMID treatment arm (Experimental): All patients enrolled received daily doses of subcutaneous injection of increased doses of anakinra starting at 0.5mg/kg/day up to a maximum 10mg/kg/day to achieve disease remission.
  Interventions: Drug: anakinra

INTERVENTIONS:
Drug: anakinra — daily injection of subcutaneous injection
  Other Names: Kineret

SUMMARY:
This study will evaluate the safety and effectiveness of anakinra (Kineret) for treating patients with neonatal-onset multisystem inflammatory disease (NOMID), also known as chronic infantile neurological, cutaneous and arthropathy (CINCA) syndrome. This disease can cause rash, joint deformities, brain inflammation, eye problems, and learning difficulties. Immune suppressing medicines commonly used to treat other pediatric rheumatologic diseases do not suppress NOMID symptoms and, if used long-term and in high doses, can cause harmful side effects. Anakinra, approved by The Food and Drug Administration for treating rheumatoid arthritis in adults, blocks a substance called IL-1 that may be an important factor in causing the inflammation in NOMID.

DETAILED DESCRIPTION:
This study uses the IL-1 receptor antagonist anakinra to treat children and adults with Neonatal-Onset Multisystem Inflammatory Disease (NOMID), also known as chronic infantile neurological, cutaneous and arthropathy (CINCA) syndrome. NOMID/CINCA syndrome is a rare genetic systemic auto-inflammatory disease that is characterized by a triad of symptoms, including a persistent urticaria-like skin rash, an arthropathy associated with patellar and epiphyseal osseous overgrowth, and neurological manifestations, including chronic aseptic meningitis, optic disc edema, high frequency hearing loss, and mental retardation. Spontaneous genetic mutations in the NACHT domain of CIAS1, a gene located on chromosome 1 have been recently identified in about half of the patients with NOMID/CINCA syndrome. CIAS1 encodes a protein, cryopyrin that is associated with up-regulation of IL-1 production in vitro, which has formed the rationale to target the IL-1 pathway in children with NOMID. During an up to 3- week enrollment period before initiating therapy, we will collect self/parent reported daily diary data and serological samples on up to 3 occasions one week apart, to determine baseline disease activity. These data may be gathered by collaborating centers. At the end of the observation period, patients will be admitted to the NIH for a standardized clinical evaluation and initiation of treatment with anakinra administered at 1 mg/kg/day by regular daily subcutaneous injections. If patients do not fulfill improvement criteria at 1 month, the dose will be escalated between 0.5 and 1 mg/kg/day increments to obtain inflammatory remission. An initial withdrawal study in a subset of 11 patients was performed. The clinical improvement at 3-4 months and the change in serum amyloid A levels (SAA) (a sensitive inflammatory marker) from before treatment to 3-4 months post treatment, and drug safety are the primary clinical outcomes of this study. To assess long-term safety and efficacy, all patients will be observed during an open ended extension phase of the study. Clinical and laboratory parameters will be used to assess safety and efficacy throughout the trial. All patients will be seen every 6 months and annually (as calculated from initiation of anakinra treatment) to further evaluate safety and long term outcomes. During the open ended extension phase of the study, patients who have residual clinical or laboratory evidence of active inflammation may have their dose increased between 0.5 and 1 mg/kg/day increments to a maximum dose of 10 mg/kg/per day to achieve clinical remission. In addition, since no data on the pharmacokinetics (PK) of anakinra in pediatric patients is available with doses exceeding 2 mg/kg/day, we plan to determine the PK of anakinra with each dose escalation.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. There is no age limitation.
2. Patients fulfill at least 2 of the following 3 clinical manifestations:

   * Typical NOMID rash
   * CNS involvement (papilledema, CSF pleocytosis, sensorineural hearing loss)
   * Typical arthropathic changes on radiograph (epiphyseal and/or patellar overgrowth.
3. Onset of manifestations of NOMID/CINCA at less than or equal to 6 months of age.
4. Stable dose of steroids, NSAIDs, DMARDs for 4 weeks prior to enrollment visit.
5. Washout period for biologics: 6 half-lives before anakinra administration for all drugs with anti TNF properties. For etanercept (6 half-lives=24 days) this calculates to drug discontinuation 3 days before enrollment into the observation period, for infliximab and adalimumab (6 half-lives=48 days) drug will be discontinued 27 before the observation period, and for thalidomide (6 half-lives=3 days) drug will be discontinued for 3 days prior to anakinra administration.
6. Patient's or legal guardian's ability and willingness to give informed consent.
7. Females of childbearing potential (young women who have had at least one menstrual period regardless of age) must have a negative urine pregnancy test at baseline prior to performance of any radiologic procedure or administration of study medication. Women of childbearing age and men able to father a child, who are sexually active, will be asked to use a form of effective birth control, including abstinence.
8. Negative PPD test using 5 T.U. intradermal testing per CDC guidelines with exception of inclusion criteria #9 below.
9. Patients with latent TB (positive PPD test) must have adequate therapy for TB initiated prior to first dose of study medication as recommended in published guidelines.

EXCLUSION CRITERIA:

1. Having received live virus vaccine during 3 months prior to baseline visit (1st visit to NIH).
2. Patients with active infections or a history of pulmonary TB infection with or without documented adequate therapy, Patients with current active TB, or recent close exposure to an individual with active TB are excluded from the study.
3. Positive testing for HIV, Hepatitis B or C known or documented at screening, enrollment or baseline visit.
4. Have a history of or concomitant diagnosis of congestive heart failure.
5. History of malignancy.
6. Recent use of IL-1 antagonist within the last three months or prior use of anti CD4 antibody.
7. Known hypersensitivity to E. coli derived products or any components of anakinra.
8. Presence of any other rheumatic disease or major chronic infectious/inflammatory/immunologic disease (e.g. inflammatory bowel disease, psoriatic arthritis, spondyloarthropathy, SLE in addition to NOMID/CINCA).
9. Presence of the following at enrollment visit: ALT or AST greater than 2.0 x upper limit of normal (ULN) of the local laboratories values, creatinine greater than 1.5 xULN, WBC less than 3.6x10(9)/l; platelet count less than 150,000 mm(3).
10. Enrollment in any other investigational clinical study or receiving an investigational agent, or has not yet completed at least 4 weeks since ending another investigational device or drug trial.
11. Subjects for whom there is concern about compliance with the protocol procedures by subject and/or parent/s and legally acceptable representative/s.
12. Lactating females or pregnant females.
13. Patients with asthma will only be included after evaluation by a pulmonary and infectious disease consultation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2003-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raphaela T Goldbach-Mansky, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
with Swedish Orphan Biovitrum Inc (SOBI)

REFERENCES:
- [Background] Feldmann J, Prieur AM, Quartier P, Berquin P, Certain S, Cortis E, Teillac-Hamel D, Fischer A, de Saint Basile G. Chronic infantile neurological cutaneous and articular syndrome is caused by mutations in CIAS1, a gene highly expressed in polymorphonuclear cells and chondrocytes. Am J Hum Genet. 2002 Jul;71(1):198-203. doi: 10.1086/341357. Epub 2002 May 24. PMID 12032915
- [Background] Hashkes PJ, Lovell DJ. Recognition of infantile-onset multisystem inflammatory disease as a unique entity. J Pediatr. 1997 Apr;130(4):513-5. No abstract available. PMID 9108844
- [Background] Hoffman HM, Mueller JL, Broide DH, Wanderer AA, Kolodner RD. Mutation of a new gene encoding a putative pyrin-like protein causes familial cold autoinflammatory syndrome and Muckle-Wells syndrome. Nat Genet. 2001 Nov;29(3):301-5. doi: 10.1038/ng756. PMID 11687797
- [Derived] Rodriguez-Smith J, Lin YC, Tsai WL, Kim H, Montealegre-Sanchez G, Chapelle D, Huang Y, Sibley CH, Gadina M, Wesley R, Bielekova B, Goldbach-Mansky R. Cerebrospinal Fluid Cytokines Correlate With Aseptic Meningitis and Blood-Brain Barrier Function in Neonatal-Onset Multisystem Inflammatory Disease: Central Nervous System Biomarkers in Neonatal-Onset Multisystem Inflammatory Disease Correlate With Central Nervous System Inflammation. Arthritis Rheumatol. 2017 Jun;69(6):1325-1336. doi: 10.1002/art.40055. Epub 2017 May 10. PMID 28118536
- [Derived] Kullenberg T, Lofqvist M, Leinonen M, Goldbach-Mansky R, Olivecrona H. Long-term safety profile of anakinra in patients with severe cryopyrin-associated periodic syndromes. Rheumatology (Oxford). 2016 Aug;55(8):1499-506. doi: 10.1093/rheumatology/kew208. Epub 2016 May 3. PMID 27143789
- [Derived] Chang Z, Spong CY, Jesus AA, Davis MA, Plass N, Stone DL, Chapelle D, Hoffmann P, Kastner DL, Barron K, Goldbach-Mansky RT, Stratton P. Anakinra use during pregnancy in patients with cryopyrin-associated periodic syndromes (CAPS). Arthritis Rheumatol. 2014 Nov;66(11):3227-32. doi: 10.1002/art.38811. PMID 25223501
- [Derived] Sibley CH, Plass N, Snow J, Wiggs EA, Brewer CC, King KA, Zalewski C, Kim HJ, Bishop R, Hill S, Paul SM, Kicker P, Phillips Z, Dolan JG, Widemann B, Jayaprakash N, Pucino F, Stone DL, Chapelle D, Snyder C, Butman JA, Wesley R, Goldbach-Mansky R. Sustained response and prevention of damage progression in patients with neonatal-onset multisystem inflammatory disease treated with anakinra: a cohort study to determine three- and five-year outcomes. Arthritis Rheum. 2012 Jul;64(7):2375-86. doi: 10.1002/art.34409. PMID 22294344
- [Derived] Goldbach-Mansky R, Dailey NJ, Canna SW, Gelabert A, Jones J, Rubin BI, Kim HJ, Brewer C, Zalewski C, Wiggs E, Hill S, Turner ML, Karp BI, Aksentijevich I, Pucino F, Penzak SR, Haverkamp MH, Stein L, Adams BS, Moore TL, Fuhlbrigge RC, Shaham B, Jarvis JN, O'Neil K, Vehe RK, Beitz LO, Gardner G, Hannan WP, Warren RW, Horn W, Cole JL, Paul SM, Hawkins PN, Pham TH, Snyder C, Wesley RA, Hoffmann SC, Holland SM, Butman JA, Kastner DL. Neonatal-onset multisystem inflammatory disease responsive to interleukin-1beta inhibition. N Engl J Med. 2006 Aug 10;355(6):581-92. doi: 10.1056/NEJMoa055137. PMID 16899778

RESULTS

PARTICIPANT FLOW:
Groups:
- NOMID: Patients who met the criteria for NOMID and treated with escalating doses of anakinra 1-5 mg/kg/day to achieve laboratory and organ inflammation remission.
Period: Overall Study
Arm/Group | NOMID
Started | 43
Completed | 41
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | NOMID
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 36
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 29
  More than one race | 1
  Unknown or Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: Diary Symptom Sum Score (DSSS) (Fever, Rash, Joint Pain, Vomiting, and Headaches)
Description: "The severity of the main symptoms of the disease were scored on a scale from 0 (no symptoms) to 4 (highest severity) on a daily basis using a diary. Five key symptoms were included in the primary variable DSSS: fever, headache, rash, joint pain, and vomiting. Each of the diary variables was evaluated as a mean value for a period preceding the visits. The baseline value was the mean value of the 5-30 last days before the first dose of Kineret. For the subsequent visits, the mean value of the last 30 days with data before each visit was used as the response variable."
Time Frame: Baseline
Population: Patients started at 1mg/kg by daily subcutaneous injection. Stepwise dose increases of 0.5-1 mg/kg/day per injection were made as frequently as every 2 weeks to achieve laboratory and organ inflammation remission. Data reported is on 26 patients who completed their 3 year assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NOMID
Number analyzed (Participants) | 26
units on a scale | 0.75741904 (0.08370955)

2. Primary Outcome: Diary Symptom Sum Score (DSSS) (Fever, Rash, Joint Pain, Vomiting, and Headaches)
Description: as for outcome 1
Time Frame: 36 months
Population: Patients started at 1mg/kg by daily subcutaneous injection. Stepwise dose increases of 0.5-1 mg/kg per injection were made as frequently as every 2 weeks up to 4.5 mg/kg/day to achieve laboratory and organ inflammation remission. Data reported is on 26 patients who completed their 3 year assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NOMID
Number analyzed (Participants) | 26
units on a scale | 0.08704545 (0.02470396)

3. Primary Outcome: Diary Symptom Sum Score (DSSS) (Fever, Rash, Joint Pain, Vomiting, and Headaches)
Description: as for outcome 1
Time Frame: 60 months
Population: Patients started at 1mg/kg by daily subcutaneous injection. Stepwise dose increases of 0.5-1 mg/kg per injection were made as frequently as every 2 weeks up to 5 mg/kg/day to achieve laboratory and organ inflammation remission. Data reported is on 20 patients who completed their 5 year assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NOMID
Number analyzed (Participants) | 20
units on a scale | 0.10768421 (0.04158048)

4. Primary Outcome: Patient / Parent Global Score of Overall Disease Activity
Description: Visual analog assessment of how arthritis affects the patient as rated by the patient themselves or parent. Measured on scale from very well (0 mm) to very poor (100 mm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NOMID
Number analyzed (Participants) | 26
units on a scale | 40.22381 (4.6242215)

5. Primary Outcome: Patient / Parent Global Score of Overall Disease Activity
Description: as for outcome 4
Time Frame: 36 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NOMID
Number analyzed (Participants) | 26
units on a scale | 8.1923077 (2.7291978)

6. Primary Outcome: Patient / Parent Global Score of Overall Disease Activity
Description: as for outcome 4
Time Frame: 60 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NOMID
Number analyzed (Participants) | 20
units on a scale | 11.1 (3.6322025)

7. Primary Outcome: Parent /Patient Pain Rating
Description: Visual analog assessment of how much pain the patient experienced in past week due to illness as rated by the patient themselves or parent. Measured on scale from no pain (0 mm) to very severe pain (100 mm).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NOMID
Number analyzed (Participants) | 26
units on a scale | 41.22381 (4.9988185)

8. Primary Outcome: Parent /Patient Pain Rating
Description: as for outcome 7
Time Frame: 36 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NOMID
Number analyzed (Participants) | 26
units on a scale | 8.9423077 (2.892075)

9. Primary Outcome: Parent /Patient Pain Rating
Description: as for outcome 7
Time Frame: 60 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NOMID
Number analyzed (Participants) | 20
units on a scale | 9.8525 (3.1635745)

10. Primary Outcome: Childhood Health Assessment Questionnaire (CHAQ)
Description: Patient self-assessment (or parent assessment) for how illness affects ability to function in daily life. Includes overall score, overall pain rating, overall global evaluation, subcategories for dressing and grooming, arising, eating, walking, hygiene, reach, grip, and activities. Measured on scale of 0-3 from 'Without any difficulty' (0) to 'Unable to do' (3).
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NOMID
Number analyzed (Participants) | 26
units on a scale | 1.1051429 (0.21122155)

11. Primary Outcome: Childhood Health Assessment Questionnaire (CHAQ)
Description: Patient self-assessment (or parent assessment) for how illness affects ability to function in daily life. Includes overall score, overall pain rating, overall global evaluation, subcategories for dressing and grooming, arising, eating, walking, hygiene, reach, grip, and activities.Measured on scale of 0-3 from 'Without any difficulty' (0) to 'Unable to do' (3).
Time Frame: 36 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NOMID
Number analyzed (Participants) | 26
units on a scale | 0.66346154 (0.15898857)

12. Primary Outcome: Childhood Health Assessment Questionnaire (CHAQ)
Description: as for outcome 10
Time Frame: 60 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NOMID
Number analyzed (Participants) | 20
units on a scale | 0.590625 (0.180202)

13. Primary Outcome: Serum Amyloid A (SAA) Measurement
Description: Serum Amyloid A is an inflammatory marker for NOMID measured using Rapid Automated Enzyme Immunoassay. Normal SAA values were defined as ≤ 10 mg/liter.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/liter
Arm/Group | NOMID
Number analyzed (Participants) | 26
mg/liter | 220.28077 (38.27684)

14. Primary Outcome: Serum Amyloid A (SAA) Measurement
Description: as for outcome 13
Time Frame: 36 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/liter
Arm/Group | NOMID
Number analyzed (Participants) | 26
mg/liter | 22.333333 (7.5122284)

15. Primary Outcome: Serum Amyloid A (SAA) Measurement
Description: as for outcome 13
Time Frame: 60 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/liter
Arm/Group | NOMID
Number analyzed (Participants) | 20
mg/liter | 21.3125 (11.586169)

16. Primary Outcome: C-reactive Protein (CRP) Measurement
Description: C-reactive protein (CRP) is an inflammatory marker for NOMID. Systemic inflammatory remission was defined as a normal CRP level (≤0.5mg/dl). Analyzed at the NIH Clinical Center Laboratory.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | NOMID
Number analyzed (Participants) | 26
mg/dl | 57.703077 (7.2213655)

17. Primary Outcome: C-reactive Protein (CRP) Measurement
Description: as for outcome 16
Time Frame: 36 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | NOMID
Number analyzed (Participants) | 26
mg/dl | 8.7511538 (2.2674947)

18. Primary Outcome: C-reactive Protein (CRP) Measurement
Description: as for outcome 16
Time Frame: 60 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | NOMID
Number analyzed (Participants) | 20
mg/dl | 6.0585 (2.3462251)

19. Primary Outcome: Erythrocyte Sedimentation Rate (ESR) Measurement
Description: Erythrocyte Sedimentation Rate (ESR) is an inflammatory marker for NOMID. Normal ESR values are defined as ≤ 25 mm/hour. Analyzed at the NIH Clinical Center Laboratory.
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | NOMID
Number analyzed (Participants) | 26
mm/hour | 56.923077 (6.3138244)

20. Primary Outcome: Erythrocyte Sedimentation Rate (ESR) Measurement
Description: as for outcome 19
Time Frame: 36 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | NOMID
Number analyzed (Participants) | 26
mm/hour | 11.576923 (1.3222045)

21. Primary Outcome: Erythrocyte Sedimentation Rate (ESR) Measurement
Description: as for outcome 19
Time Frame: 60 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | NOMID
Number analyzed (Participants) | 20
mm/hour | 11.35 (2.4355103)

ADVERSE EVENTS:
Arm/Group | NOMID
Serious Adverse Events (participants affected / at risk) | 18/43
Other Adverse Events (participants affected / at risk) | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NOMID (N=43)
hospital admission for cardiac catheterization (Cardiac disorders) | 1
Uveitis (Eye disorders) | 1
diarrhea (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
vomiting (Gastrointestinal disorders) | 1
Cytokine release syndrome (Immune system disorders) | 1
Acute Tonsillitis/tooth abscess (Infections and infestations) | 1
Appendicitis (Infections and infestations) | 1
Arthritis (Infections and infestations) | 1
Cellulitis Right lower extremity (Infections and infestations) | 1
Left cervical lymphadenitis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 2
Meningitis (Infections and infestations) | 1
Pneumonitis (Infections and infestations) | 1
Right ankle cellulitis (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Metabolic toxicity (Metabolism and nutrition disorders) | 1
generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Pain (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 5
Meningitis (Nervous system disorders) | 1
Pain (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Renal calculi (Renal and urinary disorders) | 1
Double Mastectomy (Reproductive system and breast disorders) | 1
Low grade focal ductal carcinoma in-situ of left breast (Reproductive system and breast disorders) | 1
Right breast inflammation post surgery (Reproductive system and breast disorders) | 1
Right breast scar/fibrotic tissue excised from inplant capsule (Reproductive system and breast disorders) | 1
Hospitalized for Rash (Skin and subcutaneous tissue disorders) | 1
Bilateral Capsulectomy with permenant implants (Surgical and medical procedures) | 1
L ureter stent placed (Surgical and medical procedures) | 1
Left renal stent removal (Surgical and medical procedures) | 1
Lithotripsy (Surgical and medical procedures) | 1
Post-Surgery Pneumonia (Surgical and medical procedures) | 1
Suicidal ideation (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NOMID (N=43)
Angiodema Right ring finger (Cardiac disorders) | 1
Chest wall pain (Cardiac disorders) | 4
Hypertension (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Vasovagal reaction (Cardiac disorders) | 2
ear drainage (Ear and labyrinth disorders) | 1
ear pain (Ear and labyrinth disorders) | 1
Hearing impaired (Ear and labyrinth disorders) | 2
Tinnitus (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
weight gain (Endocrine disorders) | 2
Conjunctivitis (Eye disorders) | 16
Dry eye (Eye disorders) | 1
Eye infection (Eye disorders) | 1
eye inflammation (left) (Eye disorders) | 1
Eye pain (Eye disorders) | 4
eye throbbing (Eye disorders) | 1
foreign body in eye (Eye disorders) | 1
Glaucoma (Eye disorders) | 1
hemmorage in eye (Eye disorders) | 1
itchy eyes (Eye disorders) | 1
Nystagmus (Eye disorders) | 2
Pain in extremity (Eye disorders) | 1
sty on left eye (Eye disorders) | 1
vision - eye twitch (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 7
Alanine aminotransferase increased (Gastrointestinal disorders) | 2
Anorexia (Gastrointestinal disorders) | 1
Aspartate aminotransferase increased (Gastrointestinal disorders) | 1
canker sore (Gastrointestinal disorders) | 1
Cold Sore on Gums (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 10
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 6
Gastrointestinal pain (Gastrointestinal disorders) | 6
Increased Liver Enzymes (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 6
Uveitis (Gastrointestinal disorders) | 1
vomiting (Gastrointestinal disorders) | 9
Weight loss (Gastrointestinal disorders) | 1
Disease Flare (General disorders) | 1
Fatigue (General disorders) | 7
Flare Symptoms (pt had 1 week of no anakinra) (General disorders) | 1
Flare, ran out of anakinra (General disorders) | 1
Insomnia (General disorders) | 7
Irritability (General disorders) | 1
Malaise (General disorders) | 2
NOMID Flare (General disorders) | 1
bicarbonate (Blood and lymphatic system disorders) | 1
blood / Bone Marrow - Other - elevated Hematocrit (Blood and lymphatic system disorders) | 1
blood / Bone Marrow - Other - eosinophilia (Blood and lymphatic system disorders) | 2
blood / Bone Marrow - Other - low reticulocyte count (Blood and lymphatic system disorders) | 1
Blood bilirubin increased (Blood and lymphatic system disorders) | 1
Bruising (Blood and lymphatic system disorders) | 4
Epistaxis (Blood and lymphatic system disorders) | 4
hemoglobin (Blood and lymphatic system disorders) | 1
Hypomagnesemia (Blood and lymphatic system disorders) | 1
Hyponatremia (Blood and lymphatic system disorders) | 1
Proteinuria (Blood and lymphatic system disorders) | 1
Transient elevation of LFT's (Blood and lymphatic system disorders) | 1
Allergic reaction (Immune system disorders) | 2
Allergic rhinitis (Immune system disorders) | 1
Allergic rhinitis (Infections and infestations) | 3
Blastocystis Hominis Infection (Infections and infestations) | 1
bowel abcess (Infections and infestations) | 1
Bronchial infection (Infections and infestations) | 5
Candida on palms and soles of feet bilaterally (Infections and infestations) | 1
C-Diff Recurrence (Infections and infestations) | 1
Chest Infection (?Pneumonia) (Infections and infestations) | 1
Chest wall pain (Infections and infestations) | 1
Chills (Infections and infestations) | 1
Conjunctivitis (Infections and infestations) | 4
Croup (Infections and infestations) | 1
ear drainage (Infections and infestations) | 1
Ear pain (Infections and infestations) | 1
Eczema / Atopic Dermatitis (Infections and infestations) | 1
External ear inflammation (Infections and infestations) | 14
Fever (Infections and infestations) | 16
Flu like symptoms (Infections and infestations) | 15
Folliculitis - L-Groin (Infections and infestations) | 1
G Tube Infection (Infections and infestations) | 1
Gastritis (Infections and infestations) | 7
Gastrointestinal pain (Infections and infestations) | 1
Hand-Foot-Mouth Disease (Infections and infestations) | 1
Headache (Infections and infestations) | 1
Hearing impaired (Infections and infestations) | 2
Hypopyon - Left eye (Infections and infestations) | 1
infected finger (Infections and infestations) | 1
infection without Neutropenia (Infections and infestations) | 1
infection without Neutropenia - (yeast) (Infections and infestations) | 1
infection without Neutropenia - Left arm thrombophlebitis (Infections and infestations) | 1
infection without Neutropenia - tonsillitis with sore throat (Infections and infestations) | 1
infection without Neutropenia (tooth abcess) (Infections and infestations) | 1
itchy (Infections and infestations) | 1
Lice (Infections and infestations) | 1
Lung infection (Infections and infestations) | 3
Mouth Infection (Infections and infestations) | 1
mouth sores (Infections and infestations) | 1
Nasal congestion (Infections and infestations) | 9
Oral Ulcer (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 2
Otitis media (Infections and infestations) | 10
Pharyngitis (Infections and infestations) | 3
Pneumonitis (Infections and infestations) | 1
R ear D/C (Infections and infestations) | 1
Red & burning sensation on bottom of feet (Infections and infestations) | 1
ringworm (Infections and infestations) | 1
Rotaviral Infection (Infections and infestations) | 1
RSV (Resp. Syncytial Virus) (Infections and infestations) | 1
RSV infection (Infections and infestations) | 1
Scalp Lesion (? Tinea capitis) (Infections and infestations) | 1
scarlett fever (Infections and infestations) | 1
Shingles (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 15
Skin infection (Infections and infestations) | 1
sore throat (Infections and infestations) | 10
Strep throat (Infections and infestations) | 2
strep throat (2x) (Infections and infestations) | 1
Stye (Infections and infestations) | 1
Throat infection (Infections and infestations) | 1
Tooth infection (?abscess) (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 19
Urinary tract infection (Infections and infestations) | 4
Urinary tract pain (Infections and infestations) | 5
Viral Illness (Infections and infestations) | 2
Viral Illness Dehydration (Infections and infestations) | 1
Viral Infection (Infections and infestations) | 4
Viral Infection Fever, Lethargy (Infections and infestations) | 1
Vision loss (Infections and infestations) | 1
yeast infection (Infections and infestations) | 1
Auto Accident (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 7
Physical Assault (Injury, poisoning and procedural complications) | 1
CPK increased (Investigations) | 1
Weight gain (Metabolism and nutrition disorders) | 1
Anxiety (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 16
Back pain (Musculoskeletal and connective tissue disorders) | 7
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1
Conjunctivitis (Musculoskeletal and connective tissue disorders) | 1
Dysmenorrhea (Musculoskeletal and connective tissue disorders) | 1
Edema limbs (Musculoskeletal and connective tissue disorders) | 1
Fatigue (Musculoskeletal and connective tissue disorders) | 5
Flu like symptoms (Musculoskeletal and connective tissue disorders) | 2
Fracture (Musculoskeletal and connective tissue disorders) | 3
Gait disturbance (Musculoskeletal and connective tissue disorders) | 4
Malaise (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3
Myositis (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 7
Osgood-Schlatter (Musculoskeletal and connective tissue disorders) | 1
pain (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 14
restless leg syndrome (Musculoskeletal and connective tissue disorders) | 1
S/P L Knee growth plate fixation/fever thematoma (Musculoskeletal and connective tissue disorders) | 1
A.D.D. (Nervous system disorders) | 1
Allergic reaction (Nervous system disorders) | 1
Anxiety (Nervous system disorders) | 1
Blurred vision (Nervous system disorders) | 2
carpal tunnel - right (Nervous system disorders) | 1
cerebrospinal fluid leakage (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
External ear pain (Nervous system disorders) | 1
Fever (Nervous system disorders) | 1
Generalized muscle weakness (Nervous system disorders) | 1
Glaucoma (Nervous system disorders) | 1
Headache (Nervous system disorders) | 23
Hearing impaired (Nervous system disorders) | 3
Hoarseness (Nervous system disorders) | 1
Nausea (Nervous system disorders) | 1
Neck pain (Nervous system disorders) | 1
Pain in extremity (Nervous system disorders) | 1
Paresthesia of R hand suggestive of carpel tunnel (Nervous system disorders) | 1
Saccadic Pursuit Neuropathy - Cranial (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Uveitis (Nervous system disorders) | 1
Vertigo (Nervous system disorders) | 3
vomiting (Nervous system disorders) | 1
Bladder infection (Renal and urinary disorders) | 2
Catheter related infection (Renal and urinary disorders) | 1
Flank pain (Renal and urinary disorders) | 1
glucosuria (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Ketonuria (Renal and urinary disorders) | 1
metabolic (elevated BUN) (Renal and urinary disorders) | 1
metabolic / Laboratory - Other - elevated Blood Urea Nitrogen (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal calculi (Renal and urinary disorders) | 2
Renal colic (Renal and urinary disorders) | 1
Upper respiratory infection (Renal and urinary disorders) | 2
Urinary incontinence (Renal and urinary disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 3
Urinary tract pain (Renal and urinary disorders) | 2
Breakthrough bleeding (menstrual) (Reproductive system and breast disorders) | 1
Phantom pain of breats bilateraly (Reproductive system and breast disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Gait disturbance (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 1
Allergic reaction (Skin and subcutaneous tissue disorders) | 2
bug bite (Skin and subcutaneous tissue disorders) | 1
cyst on Right cheek (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3
Eczema (contact dermatitis) (Skin and subcutaneous tissue disorders) | 1
eczematous reaction to injection (Skin and subcutaneous tissue disorders) | 1
Erythema Left Foot (Skin and subcutaneous tissue disorders) | 1
eye swollen (Skin and subcutaneous tissue disorders) | 1
fungal rash (Skin and subcutaneous tissue disorders) | 1
hive (Skin and subcutaneous tissue disorders) | 1
hives (Skin and subcutaneous tissue disorders) | 1
Hot/diaphoretic in summer months - rash at beltline (Skin and subcutaneous tissue disorders) | 1
Ingrown toenail (Skin and subcutaneous tissue disorders) | 1
Injection site reaction (Skin and subcutaneous tissue disorders) | 10
Intermittent rash on body (Skin and subcutaneous tissue disorders) | 1
lesion on scrotum (Skin and subcutaneous tissue disorders) | 1
Oral Ulcers (Skin and subcutaneous tissue disorders) | 2
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1
Penile pain (Skin and subcutaneous tissue disorders) | 1
Perineal pain (Skin and subcutaneous tissue disorders) | 1
R. 2nd toenail injury with ingrown nail (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 13
Rash - (contact dermatitis) (Skin and subcutaneous tissue disorders) | 1
Rash - adhesive (IV site) (Skin and subcutaneous tissue disorders) | 1
Rash - Bugbite - R ear (Skin and subcutaneous tissue disorders) | 1
Rash - Lichenified rash on glutial crack (Skin and subcutaneous tissue disorders) | 1
Rash - Reaction to U-bag (Skin and subcutaneous tissue disorders) | 1
Rash (viral infection) (Skin and subcutaneous tissue disorders) | 1
rash / desquamation (Skin and subcutaneous tissue disorders) | 1
Rash arms, trunk, legs (Skin and subcutaneous tissue disorders) | 1
Rash on Arms (Skin and subcutaneous tissue disorders) | 1
Rash on Right Leg (Skin and subcutaneous tissue disorders) | 1
rashes (Skin and subcutaneous tissue disorders) | 1
red cheeks (Skin and subcutaneous tissue disorders) | 1
Red Dots (Skin and subcutaneous tissue disorders) | 1
red dots - rash (Skin and subcutaneous tissue disorders) | 1
Red Dots on Arm (Skin and subcutaneous tissue disorders) | 1
Skin infection (Skin and subcutaneous tissue disorders) | 1
Cesarean Section (Surgical and medical procedures) | 1
Dental Surgery Outpatient (Surgical and medical procedures) | 1
Elective L cochlear implant surgery (Surgical and medical procedures) | 1
Elective Osteotomy (Surgical and medical procedures) | 1
Endoscopy to replace G Tube (Surgical and medical procedures) | 1
eye surgery (Surgical and medical procedures) | 1
hand surgery - carpal tunnel (Surgical and medical procedures) | 1
Kidney Stent removal (Surgical and medical procedures) | 1
Lithotripsy/stent removed (Surgical and medical procedures) | 1
Placement of BMT (tubes) (Surgical and medical procedures) | 1
staples in knee (surgery) (Surgical and medical procedures) | 1
Surgery Adenoidectomy, Placement of bilateral myringotomy tubes (Surgical and medical procedures) | 1
surgery for cyst removal (Surgical and medical procedures) | 1
surgery on right knee (Surgical and medical procedures) | 1
surgery on wrist (Surgical and medical procedures) | 1
Tonsillectomy (Surgical and medical procedures) | 1
Ureteral stent for renal calculi - Right kidney (Surgical and medical procedures) | 1
Wisdom Teeth Extraction (Surgical and medical procedures) | 1
hypertension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Data reported is on 26 patients who completed their 3 year assessment and 20 of these patients also completed their 5 year assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes